CLINICAL TRIAL: NCT01374568
Title: Changes in Bone Turnover With Increased Incretin Hormone Exposure (UAB Diabetes Research and Training Center Pilot and Feasibility Study)
Brief Title: Changes in Bone Turnover With Increased Incretin Hormone Exposure
Acronym: DRTC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed by sponsor. Funding ended.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amy H. Warriner, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UAB F100317002
Record Dates: First submitted 2011-06-10; First posted 2011-06-16 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; sitagliptin; Januvia
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sitagliptin (Active Comparator): Sitagliptin
  Interventions: Drug: sitagliptin
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: sitagliptin — sitagliptin 100mg daily
  Other Names: Januvia
  Arms: sitagliptin
Other: Placebo — 1 pill daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the use of sitagliptin increases bone formation and reduces bone turnover in postmenopausal women with type 2 diabetes.

DETAILED DESCRIPTION:
Patients with Type 2 Diabetes Mellitus (T2DM) are at an increased risk of fracture, despite having bone mineral density (BMD) similar to age and sex matched cohorts. Recent studies have indicated that changes in incretin (INtestinal seCRETion of INsulin) hormones in the setting of T2DM may play a role in bone metabolism. Two of these incretin hormones, gastric inhibitory polypeptide (GIP) and glucagon-like peptide-1 (GLP-1), have been shown to be involved in bone turnover regulation, in addition to their effect in increasing insulin secretion and decreasing glucagon secretion in a glucose-dependent manner. In addition, the rise in glucagon-like peptide-2 (GLP-2) in the postprandial state has been found to have a direct effect on reduced bone resorption in a non-fasting state and treatment with GLP-2 improved BMD in postmenopausal women. Due to their glucose lowering effects, incretins have been a therapeutic target for the treatment of T2DM through GLP-1 receptor analogs or inhibition of incretin metabolism via dipeptidyl peptidase 4 (DPP-4) inhibitors (i.e. sitagliptin). Inhibition of DPP-4 leads to an approximate doubling of GLP-1 and GIP levels but also leads to reduced breakdown of GLP-2.

Less is known about the effect of incretin-directed therapies, specifically sitagliptin, and bone metabolism. To our knowledge, two studies have looked at the direct effects of currently available incretin-directed therapies on bone metabolism. Exenatide (a GLP-1 analog) treatment of insulin resistant and type 2 diabetic rats resulted in osteogenic effects with increased osteocalcin levels following treatment. In a study of female non-diabetic Sprague-Dawley rats treated with pioglitazone, rosiglitazone, sitagliptin, vs. placebo, no significant change in bone mineral density was seen in the sitagliptin or placebo treated rats (compared to significant loss of bone mineral density in the TZD groups). Even fewer published studies are available evaluating changes in bone metabolism with the use of incretin hormones in humans. The majority of the human studies have been completed with GLP-2. These studies show a dose-dependent effect of GLP-2 on bone resorption and, preliminarily, show improved bone mineral density in postmenopausal women treated with GLP-2. However, the changes in incretin activity vary in persons with glucose intolerance and T2DM. Therefore, it is important to understand the potential effects of these medications on bone metabolism in persons prescribed these medications for treatment of their T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (as defined by age >55 years old or amenorrhea for >1years)
* Type 2 DM currently not on diabetes-specific medication(s) or treated with monotherapy of metformin or a sulfonylurea. Patients treated with insulin monotherapy will also be eligible if the total daily dose of insulin is <10units.
* Hemoglobin A1c (HbA1c) of 6.5-9.0%

Exclusion Criteria:

* Use of an incretin mimetic (i.e. exenatide), a DPP-4 inhibitor (i.e. sitagliptin, saxagliptin), a thiazolidinedione, or oral glucocorticoids in the 6 months prior to the study will not be eligible
* Known osteoporosis or patients treated with an osteoporosis-specific medication (bisphosphonate, teriparatide) or estrogen (including Selective Estrogen Receptor Modulators (SERMs)) or those who anticipate imminent treatment with one of these medications will be excluded from the study
* Chronic kidney disease (calculated GFR <30 ml/min) or a disease known to affect bone turnover (i.e. Paget Disease, Osteogenesis Imperfecta, HIV) will be excluded from the study.
* History of pancreatitis

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Warriner, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women with diabetes mellitus on no medications or metformin treatment alone were recruited from an outpatient clinic setting.
Pre-assignment Details: Potential participants completed a screening visit to ensure all study inclusion criteria were met. If on metformin at the screening visit, the metformin was discontinued. Potential participants presented 1 month later for the baseline visit and for randomization.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 2 | 3
Completed | 2 | 1
Not Completed | 0 | 2
Not completed — Lab unable to analyze BTM | 0 | 2

BASELINE CHARACTERISTICS:
Population: 6 patients were screened. 1 patient did not return for baseline visit. 5 patients were provided study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Median (Standard Deviation); unit: years] | 57.5 (6.5) | 61.0 (8.3) | 61.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
Systolic Blood Pressure [Median (Standard Deviation); unit: mmHg] | 119 (11.0) | 130 (10.0) | 130 (12.4)
Diastolic Blood Pressure [Median (Standard Deviation); unit: mmHg] | 82 (8) | 78 (6.2) | 78 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Bone Turnover in Subjects Treated With Sitagliptin When Compared to Those Treated With Placebo.
Description: Bone turnover assessed using change in TRACP5b over 8 weeks of treatment.
Time Frame: 8 weeks
Population: The difference between the bone turnover markers TRACP5b from baseline to end of study were calculated for treatment and placebo groups. Serum samples were not available for one placebo participant at baseline and for one placebo patient at end of study. As a result we were unable to analyze the 2 participants with missing data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 2 | 1
U/L | -0.25 (0.07) | 0.30 (0)

2. Primary Outcome: Bone Turnover in Subjects Treated With Sitagliptin When Compared to Those Treated With Placebo
Description: Bone turnover assessed using change in bone-specific alkaline phosphatase (BAP) over 8 weeks of treatment.
Time Frame: 8 WEEKS
Population: The difference between the bone turnover markers bone alkaline phosphatase (BAP) from baseline to end of study were calculated for treatment and placebo groups. Serum samples were not available for one placebo participant at baseline and for one placebo patient at end of study.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 2 | 1
mg/L | 0.05 (1.34) | 0 (0)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Two participants not analyzed due missing BTM at different time points. Statistician unable to include missing data due to small enrollment numbers.
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

LIMITATIONS AND CAVEATS:
Study was closed due to end of funding prior to recruitment of target participants. Small participant number limits data analysis. We were unable to obtain additional funding to complete the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No